CLINICAL TRIAL: NCT02720055
Title: Routine Exercises and Either a Psychological (Therapy-based) or a Placebo (Informational) Intervention Workbook After Distal Radius Fracture: A Double Blind Randomised Control Trial.
Brief Title: Rehabilitation Workbook After Wrist Fracture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/0037
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2016-03

CONDITIONS: Fractures, Bone
Keywords: Distal Radius Fracture; Outcomes; Psychological Intervention
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological Workbook (Experimental): Psychological work book containing information and activities aimed at improving outcomes.
  Interventions: Other: Psychological workbook
- Basic information workbook (Active Comparator): Basic information which represents current practice
  Interventions: Other: Basic information workbook

INTERVENTIONS:
Other: Psychological workbook
  Arms: Psychological Workbook
Other: Basic information workbook — Basic rehabilitation information that represents current practice.
  Arms: Basic information workbook

SUMMARY:
A randomised controlled trial to compare two different rehabilitation work books used in patients with wrist fracture.

DETAILED DESCRIPTION:
Participants

A total of 140 participants aged over 18 with distal radius fractures will be included in the study.

Sample Size The primary outcome used to calculate a sample size was the Disability of Arm Shoulder and Hand (DASH) Score. In a pilot study of sixty patients with distal radius fracture who were evaluated 8 weeks following fracture, the mean DASH score was 29 and the standard deviation was 19. A sample size of 126 would therefore provide power (90%) to identify true superiority of intervention workbook over current practice with a difference between the means equal to 10 (recognised minimal clinically significant difference in DASH) as significant at the 5% level (using a one sided test). We anticipate a drop out rate of 10% and will therefore aim to enrol 140 patients into the study. (70 in each arm).

Treatment and Rehabilitation Overview All patients will be routinely discharged from the Emergency Department following application of a cast or manipulation and application of a cast and followed up in the orthopaedic outpatient clinic. They will be treated operatively or in cast for 6 weeks (this treatment decision will be made on a clinical basis by the named consultant orthopaedic trauma surgeon responsible for the patient's care) before beginning mobilisation. All treatment types will be included in the study as no significant differences were seen between groups in terms of patient reported outcome or psychological scores in pilot study of 60 patients. Recruitment and randomisation will take place in the outpatient department at 2 weeks following injury. At this stage patients will be given one of the workbooks and instructed on how it should be used. Patients will not routinely be referred to physiotherapy but should individual patients develop a complication for which physiotherapy is clinically indicated they will be referred at this stage. Patients will be followed up at 6 weeks and 6 months following injury. The only deviation from normal practice in this trial will be the administration of the workbooks which patients will complete in their own time at home. In routine practice some patients would be followed up to 6 months, in this trial all patients will be.

Recruitment

Participants will be recruited from The Department of Orthopaedics Royal Infirmary Edinburgh. Initial management of patients in the Emergency Department and by orthopaedic services will be as routine and determined by clinical staff not involved in the trial. Fig 2.

The first potential contact with trail staff will be at the first orthopaedic outpatient appointment with in 2 weeks of injury. At this time all patients with distal radius fractures will be assessed clinically and with radiographs by the treating clinical team. Once it has been established that they fulfil trial inclusion criteria a member of the research team will be notified and the trial will be explained to the patient. They will be given a participant information sheet and if they are willing to take part, the research assistant will consent them to participate in the trial. The number of patients approached as part of the trial, the number that agree and the number that decline and for what reason will all be recorded, this data will be anonymised at the time of recording. Recruited patients will then be randomised to one of two arms: therapy based workbook intervention or placebo workbook intervention. All other treatment decisions will continue to be made by the treating clinical team.

Randomisation Participants will be randomised to routine rehabilitation plus psychological (therapy based) intervention workbook or routine rehabilitation plus placebo (information based) workbook group. Randomisation will be stratified based on age, gender and operative / non-operative treatment. Patients will be assigned to a group (A-H) based on these factors. See flow diagram Fig 1. In each group block randomisation will be carried out using a computer generated sequence. Block size will be at random (2, 4 or 6) and sequence of the block will also be at random.

Blinding Participants will be told we are comparing two different rehabilitation workbooks but will only see the workbook they are to use. They will not be given any details of the other workbook. Both workbooks will have the same format and front cover. Research team members involved in taking measurements in clinic will also be blinded to which workbook the participant is completing.

Psychological / placebo intervention Patients will complete a work book during their rehabilitation. This will begin following the 2 week follow up appointment. One arm will complete the 'Therapy Based Psychological Intervention Workbook'. It will provide information about their injury, treatment and expectations. It will address common misconceptions, negative illness perceptions and poor coping techniques and aim to improve self efficacy. This has been developed in collaboration with a Health Psychology PhD student at University of Strathclyde and agreed upon for use in this trial. This has been reviewed in a focus group of patients with distal radius fractures. The consensus was that the workbook was useful and informative. No objections were raised against the workbook. The other arm will complete a 'Placebo Workbook. This will contain stretching exercises but no therapy based exercises or exercises aimed at addressing illness perceptions or coping techniques. This placebo workbook represents the current standard of care in the Department of Orthopaedics, Royal Infirmary Edinburgh.

Baseline Information At 2 week follow up: Information regarding patient age, gender, post code, date of injury, history of previous fractures, mode of injury, associated injuries, neurovascular injury, open injury, level of pain (11 point Likert scale 0-10 low to high), past medical and psychiatric history, current medication, smoking and alcohol status, application for injury compensation, dependants, driving status, employment status, education status and level of sporting activity will be collected. All patients will complete a pre injury DASH score and SF-12. Base line Hospital anxiety and Depression score (HADS), Tampa scale for Kinesiophobia (TSK), Pain Catastrophising Score (PCS), General Self Efficacy score (SES), Recovery Locus of Control (RLoC) and Illness perception questionnaire - revised (IPQ-R), Imaging at this stage will include standardised plain film radiographs including antero posterior and lateral views of the wrist. (These radiographs are routine at this stage of treatment for patients out with the trial).

ELIGIBILITY:
Inclusion Criteria:

1. Isolated distal radius fracture undergoing management with manipulation and cast / cast alone / operative management.
2. Age 18 and over. No upper age limit

Exclusion Criteria:

1. Age < 18
2. Cognitive impairment preventing completion of patient reported questionnaires
3. Non English speaking
4. Temporary residents unable to attend follow-up
5. Patients lacking capacity to consent and patients who loose capacity during the trial.
6. Paediatric fractures in skeletally immature patients.
7. Presentation and recruitment > 3 weeks after injury
8. Patients with > 1 fracture at time of injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Disability of Arm Shoulder and Hand | 6 months
  Patient reported outcome measure validated for upper limb injuries.

SECONDARY OUTCOMES:
Objective wrist function | 6 months
  Wrist range of motion and grip strength
Patient satisfaction | 6 months
  11 point likert scale
Illness Perception Questionnaire - revised | 6 months
  scoring system for illness perception
Complications | 6 months
  record any complications

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Goudie, MBChB, Principal Investigator — NHS Lothian
Locations (1):
- Department of Orthopaedics, Royal Infirmary Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be anonymised